CLINICAL TRIAL: NCT03059056
Title: Pharmacokinetic Evaluation of Empagliflozin in Healthy Egyptian Volunteers Using LC-MS/MS: Compared With Other Ethnic Populations
Brief Title: Pharmacokinetic Evaluation of Empagliflozin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Bassam Mahfouz Ayoub, Lecturer of Pharmaceutical Chemistry, British University In Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YIRG-2016-01
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- pharmacokinetic evaluation (Experimental): Empagliflozin 25 mg
  Interventions: Drug: Empagliflozin 25mg

INTERVENTIONS:
Drug: Empagliflozin 25mg — Samples from six, healthy, adult, male, smoking, Egyptian volunteers (age: 22-33 years, Average weight: 77.8 kg, Average BMI: 29.2) will be collected at 0, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 h after administration of Empagliflozin 25 mg
  Other Names: Jardiance

SUMMARY:
Project PI (Principal Investigator): Dr Bassam Mahfouz Ayoub, Ph.D., Lecturer of Pharmaceutical Chemistry, The British University in Egypt.

Study Design The proposed study will consider the pharmacokinetic evaluation of empagliflozin after administration to Egyptian volunteers and the results will be compared with the other reported ethnic populations. The FDA recognizes that standard methods of defining racial subgroups are necessary to compare results across pharmacokinetic studies, and to assess potential subgroup differences. The design of the study is open labeled, randomized, one treatment, one period, single dose pharmacokinetic study.

DETAILED DESCRIPTION:
Study Design The proposed study will consider the pharmacokinetic evaluation of empagliflozin after administration to Egyptian volunteers and the results will be compared with the other reported ethnic populations. The FDA recognizes that standard methods of defining racial subgroups are necessary to compare results across pharmacokinetic studies, and to assess potential subgroup differences. The design of the study is open labeled, randomized, one treatment, one period, single dose pharmacokinetic study. The main pharmacokinetic parameters which are Cmax, Tmax, t1/2, elimination rate constant, AUC0-t and AUC0-inf, will be estimated. Fasting of all volunteers will eliminate the possible interaction from food or caffeine consumption. The pharmacokinetic parameters of empagliflozin will be studied in healthy human subjects according to the ethical regulations of World Medical Association Declaration of Helsinki (October 1996) and the International Conference of Harmonisation Tripartite Guideline for Good Clinical Practice. Written informed consent was provided (attached and signed by the six volunteers) in order to be approved by the ethics committee of the Faculty of Pharmacy, The British University in Egypt. The good health of the human subjects was confirmed by a complete medical history and physical examination. Samples from six, healthy, adult, male, smoking, Egyptian volunteers (age: 22-33 years, Average weight: 77.8 kg, Average BMI: 29.2) will be collected at 0, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 h, to be transferred to heparinized centrifuge tubes in order to be analyzed by LC-MS/MS study (developed & validated) after single oral dose administration of one Jardiance® tablet nominally containing 25 mg of empagliflozin. The blood samples (3 mL of each sample) will be centrifuged at 3000 rpm for 5 minutes, one mL of the plasma will be separated and spiked with 100 µL (equivalent to 100 ng) of internal standard working solution and then the sample preparation and LC-MS/MS determination will be applied. The main pharmacokinetic parameters of the study which are Cmax, Tmax, t1/2, elimination rate constant, AUC0-t and AUC0-inf will be estimated, using a validated excel software. Blood glucose level will be determined for all volunteers at different time intervals to monitor any hypoglycemic effect. The study will be conducted as per FDA guidelines. The development of such correlations between empagliflozin concentrations and its pharmacologic responses will enable clinicians to apply pharmacokinetic principles to actual patient situations. The evaluation of safety of the study will be based on monitoring of blood glucose level, vital signs, pulse rate, monitoring of adverse events, and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* The good health of the human subjects was confirmed by a complete medical history and physical examination.

Exclusion Criteria:

* Chronic disease

Ages: 22 Years to 33 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Cmax | 12 Hours
  The peak plasma concentration of a drug after administration
Tmax | 12 Hours
  Time to reach Cmax.
Elimination half life | 12 Hours
  The time required for the concentration of the drug to reach half of its original value.
Elimination rate constant | 12 Hours
  The rate at which a drug is removed from the body.
Area under the curve | 12 Hours
  The integral of the concentration-time curve

IPD SHARING:
Plan to Share IPD: Yes
Publication of data in a scientific journal